CLINICAL TRIAL: NCT00784225
Title: S0000B: Prevention of Cataract and Age-Related Macular Degeneration With Vitamin E and Selenium - SELECT Eye Endpoints (SEE)
Brief Title: S0000B: Vitamin E and/or Selenium in Preventing Cataract and Age-Related Macular Degeneration in Men on SELECT SWOG-S0000
Acronym: SEE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CDR0000617778; S0000B (Other: SWOG); U10CA037429 (NIH); R01EY014418 (NIH)
Record Dates: First submitted 2008-10-31; First posted 2008-11-03 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Cataract; Macular Degeneration
Keywords: cataract; advanced macular degeneration
MeSH Terms: conditions — Cataract; Macular Degeneration | interventions — Selenium; Vitamin E; alpha-Tocopherol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vitamin E + selenium placebo (Experimental): vitamin E and selenium placebo daily for 7-12 years
  Interventions: Drug: vitamin E; Drug: selenium placebo
- Selenium + vitamin E placebo (Experimental): selenium and vitamin E placebo daily for 7-12 years
  Interventions: Drug: selenium; Drug: vitamin E placebo; Drug: selenium placebo
- Vitamin E + selenium (Experimental): vitamin E and selenium placebo daily for 7-12 years
  Interventions: Drug: selenium; Drug: vitamin E
- Vitamin E placebo + selenium placebo (Placebo Comparator): vitamin E placebo and selenium placebo daily for 7-12 years
  Interventions: Drug: vitamin E placebo; Drug: selenium placebo

INTERVENTIONS:
Drug: selenium — 200 mcg daily for 7-12 years
  Other Names: L-selenomethionine
  Arms: Selenium + vitamin E placebo; Vitamin E + selenium
Drug: vitamin E — 400 IU daily by mouth for 7-12 years
  Other Names: alpha tocopherol
  Arms: Vitamin E + selenium; Vitamin E + selenium placebo
Drug: vitamin E placebo — daily for 7-12 years
  Other Names: placebo
  Arms: Selenium + vitamin E placebo; Vitamin E placebo + selenium placebo
Drug: selenium placebo — daily for 7-12 years
  Other Names: placebo
  Arms: Selenium + vitamin E placebo; Vitamin E + selenium placebo; Vitamin E placebo + selenium placebo

SUMMARY:
RATIONALE: Aging may affect a person's vision. Vitamin E and/or selenium may help prevent cataracts or age-related macular degeneration in men receiving these drugs as part of a clinical trial for the prevention of prostate cancer.

PURPOSE: This clinical trial is studying vitamin E and/or selenium to see how well they work in preventing cataract and age-related macular degeneration in men enrolled on SELECT (SWOG-S0000).

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To test whether vitamin E and/or selenium reduces the risk of visually significant age-related macular degeneration (AMD) in men enrolled on SELECT (SWOG-S0000).
* To test whether vitamin E and/or selenium reduces the risk of cataract in these participants.

Secondary

* To test whether vitamin E and/or selenium reduces the risk of advanced AMD in these participants.
* To test whether vitamin E and/or selenium reduces the risk of cataract surgery and subtypes in these participants.

OUTLINE: This is a multicenter study.

Data from medical records obtained from the participant's ophthalmologist or optometrist are reviewed. Information from these records is then used to confirm baseline reports of age-related macular degeneration (AMD) as well as 6-month and annual reports of new diagnoses of AMD and cataract (or cataract surgery) made since the start of this study. Detailed questionnaires are also obtained from the participant's ophthalmologist or optometrist to provide information about the reported AMD or cataract diagnosis (e.g., date of initial diagnosis; best-corrected visual acuity at the time of diagnosis; date when visual acuity was first noted to be 20/30 or worse [if different from the date of initial diagnosis]; pathological findings observed when AMD was first diagnosed [e.g., drusen, retinal pigment epithelial hypo/hyperpigmentation, geographic atrophy, retinal pigment epithelial detachment, subretinal neovascular membrane, or disciform scar]; pathological findings observed when visual acuity was first noted to be 20/30 or worse; date when exudative [wet] AMD was first noted; presence of other ocular abnormalities that could explain or contribute to visual loss; whether AMD or cataract, by itself, are significant enough to cause vision to be reduced to 20/30 or worse; whether laser treatment or photodynamic therapy was performed for AMD; date of cataract extraction; etiology of cataract [e.g., age-related, traumatic, congenital, inflammatory, or surgery- or steroid-induced]; and cataract type [e.g., nuclear, cortical, posterior subcapsular, or other]).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Enrolled on the Selenium and Vitamin E Prostate Cancer Prevention Trial (SELECT) SWOG-S0000
* Diagnosis of 1 of the following:

  * Age-related macular degeneration (AMD) at baseline or at follow-up
  * Cataract or a cataract extraction at follow-up (Closed for accrual as of 10/01/29)

    * Participants with a prior diagnosis of cataract at baseline followed by another cataract event (cataract diagnosis or a cataract extraction) at follow-up are not eligible
    * Participants with a prior diagnosis of cataract at baseline followed by a diagnosis of AMD at follow-up are eligible

PATIENT CHARACTERISTICS:

* See Disease Characteristics

PRIOR CONCURRENT THERAPY:

* Not applicable

Ages: 50 Years to 120 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13475 (Actual)
Dates: Start 2004-07; Primary Completion 2017-11 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Christen, ScD, Study Chair — Dana-Farber/Brigham and Women's Cancer Center
Locations (1):
- Harvard Medical School, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Goodman PJ, Tangen CM, Darke AK, Arnold KB, Hartline J, Yee M, Anderson K, Caban-Holt A, Christen WG, Cassano PA, Lance P, Klein EA, Crowley JJ, Minasian LM, Meyskens FL. Opportunities and challenges in incorporating ancillary studies into a cancer prevention randomized clinical trial. Trials. 2016 Aug 12;17:400. doi: 10.1186/s13063-016-1524-9. PMID 27519183
- [Derived] Christen WG, Glynn RJ, Gaziano JM, Darke AK, Crowley JJ, Goodman PJ, Lippman SM, Lad TE, Bearden JD, Goodman GE, Minasian LM, Thompson IM Jr, Blanke CD, Klein EA. Age-related cataract in men in the selenium and vitamin e cancer prevention trial eye endpoints study: a randomized clinical trial. JAMA Ophthalmol. 2015 Jan;133(1):17-24. doi: 10.1001/jamaophthalmol.2014.3478. PMID 25232809

RESULTS

PARTICIPANT FLOW:
Groups:
- Selenium + Vitamin E Placebo: Patients received selenium and vitamin E placebo daily for 7 - 12 years
  Selenium: 200 mcg daily for 7 - 12 years
  Vitamin E placebo: 1 pill by mouth daily for 7 - 12 years
- Selenium + Vitamin E: Patients received selenium and vitamin E daily for 7 - 12 years
  Selenium: 200 mcg 1 pill by mouth daily for 7 - 12 years
  Vitamin E: 400 IU daily by mouth for 7 - 12 years
- Vitamin E Placebo + Selenium Placebo: Patients received vitamin E placebo and selenium placebo daily for 7 - 12 years
  Vitamin E placebo:1 pill daily by mouth for 7 - 12 years
  Selenium placebo: 1 pill by mouth daily for 7 - 12 years
- Vitamin E + Selenium Placebo: Patients received vitamin E and selenium placebo daily for 7 - 12 years
  Vitamin E: 400 IU by mouth daily for 7 - 12 years
  Selenium placebo: 1 pill by mouth daily for 7 - 12 years
Period: Overall Study
Arm/Group | Selenium + Vitamin E Placebo | Selenium + Vitamin E | Vitamin E Placebo + Selenium Placebo | Vitamin E + Selenium Placebo
Started | 3375 | 3357 | 3369 | 3374
Completed | 3375 | 3357 | 3369 | 3374
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants at SELECT sites with IRB approval for SEE and who agreed to participate in SEE or were willing to be contacted about registering to SEE if they were to have an eye event were registered to AMD (13389) and Cataract (11267) portions. There was overlap between the two populations.
Groups:
- Selenium + Vitamin E Placebo: Selenium and vitamin E placebo daily for 7-12 years.
  Selenium: 200 mcg daily for 7 - 12 years
  Vitamin E placebo: 1 pill by mouth daily for 7 - 12 years
- Selenium + Vitamin E: Selenium and vitamin E daily for 7-12 years. Selenium: 200 mcg daily for 7 - 12 years
  Vitamin E: 400 IU daily by mouth for 7 - 12 years
- Vitamin E Placebo + Selenium Placebo: Vitamin E placebo and selenium placebo daily for 7-12 years.
  Vitamin E placebo: 1 pill by mouth daily for 7 - 12 years
  Selenium placebo: 1 pill by mouth daily for 7 - 12 years
- Vitamin E + Selenium Placebo: Vitamin E and selenium placebo daily for 7-12 years.
  Vitamin E: 400 IU daily by mouth for 7 - 12 years
  Selenium placebo: 1 pill by mouth daily for 7 - 12 years
- Total: Total of all reporting groups
Arm/Group | Selenium + Vitamin E Placebo | Selenium + Vitamin E | Vitamin E Placebo + Selenium Placebo | Vitamin E + Selenium Placebo | Total
Number analyzed (Participants) | 3375 | 3357 | 3369 | 3374 | 13475
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [58 to 68] | 62 [58 to 67] | 62 [58 to 67] | 62 [57 to 67] | 62 [58 to 67]
Age, Customized [Count of Participants; unit: Participants]
  50-54 years | 134 | 160 | 159 | 155 | 608
  55-64 years | 1951 | 1964 | 1959 | 2027 | 7901
  65-74 years | 1065 | 1067 | 1061 | 993 | 4186
  >=75 years | 225 | 166 | 190 | 199 | 780
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 3375 | 3357 | 3369 | 3374 | 13475
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2753 | 2756 | 2750 | 2763 | 11022
  Non-white | 622 | 601 | 619 | 611 | 2453
Education (highest level) [Count of Participants; unit: Participants]
  <= High school graduate or GED | 653 | 641 | 706 | 656 | 2656
  Some college/vocational school | 943 | 943 | 948 | 964 | 3798
  >College graduate | 1759 | 1752 | 1705 | 1738 | 6954
  Unknown/missing | 20 | 21 | 10 | 16 | 67
Cigarette smoking [Count of Participants; unit: Participants]
  Never | 1451 | 1419 | 1366 | 1457 | 5693
  Current | 248 | 278 | 319 | 268 | 1113
  Former | 1670 | 1654 | 1681 | 1642 | 6647
  Unknown | 6 | 6 | 3 | 7 | 22
Alcohol use [Count of Participants; unit: Participants]
  Rarely/never | 50 | 51 | 66 | 59 | 226
  >=1 drink/month | 3325 | 3304 | 3303 | 3314 | 13246
  Unknown | 0 | 2 | 0 | 1 | 3
Body mass index (kg/m^2) [Count of Participants; unit: Participants]
  <25 | 674 | 666 | 675 | 626 | 2641
  25-<30 | 1574 | 1607 | 1591 | 1606 | 6378
  >=30 | 1127 | 1084 | 1103 | 1142 | 4456
History of hypertension [Count of Participants; unit: Participants]
  Yes | 1339 | 1320 | 1374 | 1301 | 5334
  No | 2036 | 2037 | 1995 | 2073 | 8141
Aspirin use [Count of Participants; unit: Participants]
  Yes | 1484 | 1454 | 1505 | 1481 | 5924
  No | 1891 | 1903 | 1864 | 1893 | 7551
Statin use [Count of Participants; unit: Participants]
  Yes | 884 | 886 | 900 | 914 | 3584
  No | 2464 | 2447 | 2451 | 2434 | 9796
  Unknown | 27 | 24 | 18 | 26 | 95
History of diabetes [Count of Participants; unit: Participants]
  Yes | 353 | 348 | 380 | 339 | 1420
  No | 3022 | 3009 | 2989 | 3035 | 12055
Records sought [Count of Participants; unit: Participants] — Participants were asked to consent to participate in S0000B, which required them to complete a medical release with information about their ophthalmologic provider. Using this information, Providers were sent a form to complete describing the cataract/cataract extraction/AMD (as applicable) in detail.
  Participants
    Yes | 635 | 624 | 624 | 629 | 2512
    No | 2740 | 2733 | 2745 | 2745 | 10963
Included in cataract analysis [Count of Participants; unit: Participants]
  Yes | 2805 | 2789 | 2829 | 2844 | 11267
  No | 570 | 568 | 540 | 530 | 2208
Included in AMD analysis [Count of Participants; unit: Participants]
  Yes | 3348 | 3342 | 3355 | 3344 | 13389
  No | 27 | 15 | 14 | 30 | 86

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Visually Significant Age-related Macular Degeneration (AMD)
Description: Visually significant age-related AMD was defined as incident AMD responsible for reduction in best corrected visual acuity to 20/30 or worse(AMD 20/30)
Time Frame: Every 6 months, up to 7 years
Population: Marginal analyses were performed with arms pooled based on active vs. placebo selenium or vitamin E.
Measure: Count of Participants; unit: Participants
Groups:
- AMD: Selenium Active: Patients received selenium and either Vitamin E or vitamin E placebo daily for 7 - 12 years
  Selenium: 200 mcg daily for 7 - 12 years
  Vitamin E: 400 IU daily by mouth for 7 - 12 years
  Vitamin E placebo: 1 pill by mouth daily for 7 - 12 years
- AMD: Selenium Placebo: Patients received selenium placebo and either Vitamin E or vitamin E placebo daily for 7 - 12 years
  Selenium placebo: 1 pill by mouth daily for 7 - 12 years
  Vitamin E: 400 IU daily by mouth for 7 - 12 years
  Vitamin E placebo: 1 pill by mouth daily for 7 - 12 years
- AMD: Vitamin E Active: Patients received vitamin E and either selenium or selenium placebo daily for 7 - 12 years
  Vitamin E: 400 IU daily by mouth for 7 - 12 years
  Selenium: 200 mcg daily for 7 - 12 years
  Selenium placebo: 1 pill by mouth daily for 7 - 12 years
- AMD: Vitamin E Placebo: Patients received vitamin E placebo and either selenium or selenium placebo daily for 7 - 12 years
  Vitamin E placebo: 1 pill by mouth daily for 7 - 12 years
  Selenium: 200 mcg daily for 7 - 12 years
  Selenium placebo: 1 pill by mouth daily for 7 - 12 years
Arm/Group | AMD: Selenium Active | AMD: Selenium Placebo | AMD: Vitamin E Active | AMD: Vitamin E Placebo
Number analyzed (Participants) | 6690 | 6699 | 6686 | 6703
Participants
  AMD cases | 9 | 12 | 9 | 12
  non-AMD cases | 6681 | 6687 | 6677 | 6691
Statistical Analysis 1: Comparison: AMD: Selenium Active vs AMD: Selenium Placebo; Statistical analysis for number of participants with visually significant AMD in SEE sites during pill-taking for selenium; Test type: Superiority; p = 0.52, Regression, Cox; Cox Proportional Hazard = 0.75, 95% CI 2-sided [0.32 to 1.79]
Statistical Analysis 2: Comparison: AMD: Vitamin E Active vs AMD: Vitamin E Placebo; Statistical analysis for number of participants with visually significant AMD in SEE sites during pill-taking for vitamin E; Test type: Superiority; p = 0.51, Regression, Cox; Cox Proportional Hazard = 0.75, 95% CI 2-sided [0.31 to 1.77]

2. Primary Outcome: Number of Participants With Cataract and Best Corrected Visual-acuity of 20/30
Description: Incident cataract was defined as lens opacity diagnosed after randomization but prior to end of study, age-related in origin, and best-corrected visual acuity of 20/30 or worse attributable to the opacity.
Time Frame: Every 6 months, up to 7 years
Population: Marginal analyses were performed with arms pooled based on active vs. placebo selenium or vitamin E.
Measure: Count of Participants; unit: Participants
Groups:
- Cataract: Selenium Active: Patients received selenium and either vitamin E or vitamin E placebo daily for 7 - 12 years
  Selenium: 200 mcg daily for 7 - 12 years
  Vitamin E: 400 IU daily by mouth for 7 - 12 years
  Vitamin E placebo: 1 pill by mouth daily for 7 - 12 years
- Cataract: Selenium Placebo: Patients received selenium placebo and either vitamin E or vitamin E placebo daily for 7 - 12 years
  Selenium placebo: 1 pill by mouth daily for 7 - 12 years
  Vitamin E: 400 IU daily by mouth for 7 - 12 years
  Vitamin E placebo: 1 pill by mouth daily for 7 - 12 years
- Cataract: Vitamin E Active: Patients received vitamin E and either selenium or selenium placebo daily for 7 - 12 years
  Vitamin E: 400 IU daily by mouth for 7 - 12 years
  Selenium: 200 mcg daily for 7 - 12 years
  Selenium placebo: 1 pill by mouth daily for 7 - 12 years
- Cataract: Vitamin E Placebo: Patients received vitamin E placebo and either selenium or selenium placebo daily for 7 - 12 years
  Vitamin E placebo: 1 pill by mouth daily for 7 - 12 years
  Selenium: 200 mcg daily for 7 - 12 years
  Selenium placebo: 1 pill by mouth daily for 7 - 12 years
Arm/Group | Cataract: Selenium Active | Cataract: Selenium Placebo | Cataract: Vitamin E Active | Cataract: Vitamin E Placebo
Number analyzed (Participants) | 5594 | 5673 | 5633 | 5634
Participants
  Cataract cases | 185 | 204 | 197 | 192
  non-cataract cases | 5409 | 5469 | 5436 | 5442
Statistical Analysis 1: Comparison: Cataract: Selenium Active vs Cataract: Selenium Placebo; Test type: Superiority; p = 0.37, Regression, Cox; Cox Proportional Hazard = 0.91, 95% CI 2-sided [0.75 to 1.11]
Statistical Analysis 2: Comparison: Cataract: Vitamin E Active vs Cataract: Vitamin E Placebo; Test type: Superiority; p = 0.81, Regression, Cox; Cox Proportional Hazard = 1.02, 95% CI 2-sided [0.84 to 1.25]

3. Secondary Outcome: Number of Participants With Advanced AMD
Description: Advanced AMD was defined as the occurrence of disciform scars, or geographic atrophy or retinal pigment epithelium (RPE) detachment in either or both eyes at AMD diagnosis.
Time Frame: Every 6 months, up to 7 years
Population: Marginal analyses were performed with arms pooled based on active vs. placebo selenium or vitamin E.
Measure: Count of Participants; unit: Participants
Arm/Group | AMD: Selenium Active | AMD: Selenium Placebo | AMD: Vitamin E Active | AMD: Vitamin E Placebo
Number analyzed (Participants) | 6690 | 6699 | 6686 | 6703
Participants
  Advanced AMD cases | 10 | 4 | 7 | 7
  non-advanced AMD cases | 6680 | 6695 | 6679 | 6696
Statistical Analysis 1: Comparison: AMD: Selenium Active vs AMD: Selenium Placebo; Statistical analysis for number of participants with advanced AMD in SEE sites during pill-taking for selenium; Test type: Superiority; p = 0.12, Regression, Cox; Cox Proportional Hazard = 2.5, 95% CI 2-sided [0.79 to 7.98]
Statistical Analysis 2: Comparison: AMD: Vitamin E Active vs AMD: Vitamin E Placebo; Statistical analysis for number of participants with advanced AMD in SEE sites during pill-taking for vitamin E; Test type: Superiority; p = 0.98, Regression, Cox; Cox Proportional Hazard = 0.99, 95% CI 2-sided [0.35 to 2.82]

4. Secondary Outcome: Number of Participants Who Underwent Cataract Extraction
Description: Cataract extraction was defined as the surgical removal of an incident cataract.
Time Frame: Every 6 months, up to 7 years
Population: Marginal analyses were performed with arms pooled based on active vs. placebo selenium or vitamin E.
Measure: Count of Participants; unit: Participants
Arm/Group | Cataract: Selenium Active | Cataract: Selenium Placebo | Cataract: Vitamin E Active | Cataract: Vitamin E Placebo
Number analyzed (Participants) | 5594 | 5673 | 5633 | 5634
Participants
  Cataract extraction cases | 99 | 120 | 114 | 105
  non-cataract extraction cases | 5495 | 5553 | 5519 | 5529
Statistical Analysis 1: Comparison: Cataract: Selenium Active vs Cataract: Selenium Placebo; Test type: Superiority; p = 0.19, Regression, Cox; Cox Proportional Hazard = 0.84, 95% CI 2-sided [0.64 to 1.09]
Statistical Analysis 2: Comparison: Cataract: Vitamin E Active vs Cataract: Vitamin E Placebo; Test type: Superiority; p = 0.58, Regression, Cox; Cox Proportional Hazard = 1.08, 95% CI 2-sided [0.83 to 1.41]

ADVERSE EVENTS:
Time Frame: Every 6 months while the participant is receiving study supplements, up to 7 years
Description: There are no Adverse Events (AE) associated with this trial. All AEs were reported for the parent trial (SELECT - S0000). Included below are the AEs for the participants on this trial that were included in the primary analysis. These AEs were also reported for the parent trial.
Groups:
- Selenium + Vitamin E Placebo: Selenium + Vitamin E placebo
- Selenium + Vitamin E: Selenium + Vitamin E
- Placebo: Placebo
- Vitamin E + Selenium Placebo: Vitamin E + Selenium placebo
Arm/Group | Selenium + Vitamin E Placebo | Selenium + Vitamin E | Placebo | Vitamin E + Selenium Placebo
All-Cause Mortality (participants affected / at risk) | 151/3374 | 159/3356 | 150/3366 | 147/3374
Serious Adverse Events (participants affected / at risk) | 44/3374 | 41/3356 | 50/3366 | 45/3374
Other Adverse Events (participants affected / at risk) | 243/3374 | 243/3356 | 261/3366 | 267/3374
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Selenium + Vitamin E Placebo (N=3374) | Selenium + Vitamin E (N=3356) | Placebo (N=3366) | Vitamin E + Selenium Placebo (N=3374)
Arrhythmia, NOS (Cardiac disorders) | 1 | 1 | 0 | 0
Cardiac ischemia/infarction (Cardiac disorders) | 11 | 9 | 9 | 8
Cardiovascular-other (Cardiac disorders) | 7 | 9 | 15 | 12
Conduction abnormality/block (Cardiac disorders) | 0 | 1 | 0 | 0
LVEF decrease/CHF (Cardiac disorders) | 2 | 0 | 0 | 1
Supraventricular arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 1 | 3 | 2
Eye-other (Eye disorders) | 0 | 0 | 0 | 1
Vision,NOS (Eye disorders) | 0 | 0 | 1 | 0
GI-other (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Melena/ GI bleeding (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Constitutional symptoms-other (General disorders) | 0 | 0 | 1 | 0
Hemorrhage w/o 3-4 thrombocyt (General disorders) | 0 | 0 | 0 | 1
Reportable adverse event, NOS (General disorders) | 8 | 7 | 11 | 8
Liver-clinical (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Respiratory infect w/o neutrop (Infections and infestations) | 2 | 0 | 1 | 1
Respiratory infection, unk ANC (Infections and infestations) | 0 | 0 | 0 | 1
Surgery-hemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Weight gain (Investigations) | 0 | 0 | 1 | 0
Second primary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4 | 1 | 0
CNS hemorrhage (Nervous system disorders) | 2 | 2 | 0 | 3
Cerebrovascular ischemia (Nervous system disorders) | 2 | 4 | 1 | 4
Seizures (Nervous system disorders) | 1 | 0 | 0 | 0
Sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Emphysema/COPD (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Carotid stenosis (Vascular disorders) | 0 | 1 | 0 | 1
Peripheral arterial ischemia (Vascular disorders) | 0 | 1 | 1 | 0
Thrombosis/embolism (Vascular disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Selenium + Vitamin E Placebo (N=3374) | Selenium + Vitamin E (N=3356) | Placebo (N=3366) | Vitamin E + Selenium Placebo (N=3374)
Cardiac ischemia/infarction (Cardiac disorders) | 243 | 243 | 261 | 267

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2009-10-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT00784225/Prot_SAP_ICF_000.pdf